CLINICAL TRIAL: NCT03742167
Title: Pilot Randomized Control Trial of Telemedical Support for Paramedics in Simulated Pre-hospital Pediatric Emergencies
Brief Title: Pilot Simulation RCT of Telemedical Support for Paramedics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-37817; K23HL145126-01A1 (NIH)
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Respiratory Failure; Status Epilepticus; Status Asthmaticus; Cardiopulmonary Arrest
Keywords: Prehospital emergency care; Paramedic performance; Telemedicine; Medical control physician; Infant mannequin smulation; Pediatric life threatening illness
MeSH Terms: conditions — Respiratory Insufficiency; Status Epilepticus; Status Asthmaticus; Heart Arrest | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Live and video raters of paramedic performance are blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine (Experimental): The telemedicine arm will have 2-way audiovisual connection with a pediatric medical control physician.
  Interventions: Other: Telemedicine
- Control (No Intervention): The control arm will receive pediatric medical control physician consultation via telephone.

INTERVENTIONS:
Other: Telemedicine — The mobile, HIPAA-compliant, video-conferencing platform, Zoom Pro, will be used on tablet computers as a low-cost telemedicine platform for the intervention group. This platform uses Wi-Fi or cellular data connection for video streaming. The investigators will use the telephone communication on this platform for control scenarios, to mimic the current standard for audio-only consultation. A web-based software platform (WireCast®) will capture video recordings over a secure wireless network.
  Arms: Telemedicine

SUMMARY:
This study evaluates the impact of video communication via telemedicine on the quality of emergency care provided to children by paramedic teams supported by a remote physician in a simulated out-of-hospital setting. Half of the paramedic teams will use a video telemedicine platform for communication with a physician, while the other half will use an audio-only platform.

DETAILED DESCRIPTION:
In the United States, the current standard of pre-hospital (out-of-hospital) emergency care for children with life-threatening illnesses in the community includes remote physician medical direction for paramedics providing life-saving therapies while transporting the child to the hospital. Most pre-hospital emergency medical service (EMS) agencies use radios systems for audio communication between paramedics and physicians. This communication strategy is inherently limited as the remote physician cannot visualize the patient for accurate assessment and to direct treatment.

The purpose of this pilot study is to evaluate whether use of a 2-way audiovisual connection with a pediatric emergency medicine expert (intervention = "telemedical support") will improve the quality of care provided by paramedics to infant simulator mannequins with life-threatening illnesses. Paramedics receiving real-time telemedical support by a pediatric expert may provide better care due to decreased cognitive burden, critical action checking, protocol verification, and error correction.

Because real pediatric life-threatening illnesses are rare, high-stakes events and involve a vulnerable population (children), this pilot randomized control trial will provide early data on the efficacy of this intervention in simulated cases of pediatric medical emergencies. The primary outcome is "paramedic resuscitation performance" measured by a checklist of observable critical actions by independent reviewers during live observation and video review. The results of this study will provide important pilot data to estimate the clinical effect of this intervention and the sample size needed for a future definitive trial with children, a vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Certified paramedics from three EMS systems in the Boston metropolitan area (Boston EMS, South Shore EMS, and Lahey Medical Center EMS)
* Attending physicians and clinical fellows with expertise in pediatric emergency medicine and pediatric resuscitation from 2 pediatric referral centers (Boston Medical Center and Boston Children's Hospital)

Exclusion Criteria:

-Prehospital providers without paramedic level certification (e.g. BLS certification only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Paramedic Team Performance score | 9 months
  The paramedic team performance score is generated from a 64-item checklist of observable actions for pediatric assessment and resuscitation that are scored dichotomously (observed/not observed). The composite performance score is calculated as the number of observed actions divided by the total number of expected actions per case, and reported as a percentage of completed observed actions. This checklist is validated for simulation-based assessment of paramedic performance using three simulated cases of pediatric pre-hospital emergencies. Paramedic team performance will be rated by 1 live and 2 video raters. The final performance score for each team will be reported as an average score for all three raters.

SECONDARY OUTCOMES:
NASA Task load Index | 9 months
  This is an extensively validated measure of perceived workload of individuals. It is a multidimensional scale where individuals estimate workload during or after completing a task. It contains 7 domains (mental demand, physical demand, temporal demand, performance, effort, frustration, and anxiety) which are evaluated on a 20-point Likert scale. Study participants will complete this questionnaire immediately after completing the simulation modules.
Telemedicine Platform Usability | 9 months
  This 14-item questionnaire is a validated measure of all the usability of telehealth platforms (usefulness, ease of use, effectiveness, reliability, and satisfaction). The investigators modified this questionnaire to specifically address the usability of a prehospital telemedicine platform. Study participants will complete this questionnaire immediately after completing the simulation modules.
Error in medication choice | 9 months
  This will be any incorrect type of medication utilized by a team during each simulation resuscitation. This includes unanticipated medication choices which the study raters feel was not indicated or potentially harmful by consensus opinion. This data is collected in the paramedic performance checklist.
Error in weight-based medication dosing | 9 months
  This will include any errors in pediatric weight-based dose calculation, including errors in volume of drug administered during each simulated case. This data is collected in the paramedic performance checklist.
Equipment size error | 9 months
  This includes errors in equipment size during each simulated resuscitation. This data is collected in the paramedic performance checklist.
Equipment use errors | 9 months
  This includes errors in equipment usage (e.g. depth of endotracheal tube insertion, rate of bag-valve-mask ventilation, location of intraosseous needle insertion) during each simulated resuscitation. This data is collected in the paramedic performance checklist.
EMS protocol error | 9 months
  This will be defined as any error in offline and online EMS treatment protocols that is observed during each simulated resuscitation. This data is collected in the paramedic performance checklist.

CONTACTS AND LOCATIONS:
Overall Officials: Tehnaz Boyle, MD PhD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lammers RL, Byrwa MJ, Fales WD, Hale RA. Simulation-based assessment of paramedic pediatric resuscitation skills. Prehosp Emerg Care. 2009 Jul-Sep;13(3):345-56. doi: 10.1080/10903120802706161. PMID 19499472
- [Background] Butler L, Whitfill T, Wong AH, Gawel M, Crispino L, Auerbach M. The Impact of Telemedicine on Teamwork and Workload in Pediatric Resuscitation: A Simulation-Based, Randomized Controlled Study. Telemed J E Health. 2019 Mar;25(3):205-212. doi: 10.1089/tmj.2018.0017. Epub 2018 Jun 29. PMID 29957150
- [Background] Parmanto B, Lewis AN Jr, Graham KM, Bertolet MH. Development of the Telehealth Usability Questionnaire (TUQ). Int J Telerehabil. 2016 Jul 1;8(1):3-10. doi: 10.5195/ijt.2016.6196. eCollection 2016 Spring. PMID 27563386